CLINICAL TRIAL: NCT06346886
Title: FAITH! Hypertension App to Improve Hypertension Control and Cardiovascular Health Among African-Americans: A Decentralized Randomized Clinical Trial
Brief Title: HTN App for HTN Control and Cardiovascular Health Among African-Americans
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Miami Heart Research Institute Inc. (Unknown)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-011703
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): African American adults with uncontrolled hypertension (HTN) will be assigned to complete an 11 week guided intervention using the FAITH! HTN app.
  Interventions: Behavioral: FAITH! HTN app
- Control Group (No Intervention): African American adults with uncontrolled hypertension (HTN) will receive the standard of care of HTN management.

INTERVENTIONS:
Behavioral: FAITH! HTN app — Participants will remain in the intervention for 11 weeks. The app-based intervention is a tailored program to promote HTN self-management and knowledge through an 11-module educational video series with a focus on HTN. Participants will also be provided with at home Blood Pressure (BP) monitoring system to allow for self-tracking of BP measurements(automatically synchronized with the app). The app will include pre-post module quizzes, a tracking component for participants to input self-monitored measures (medication adherence, diet, physical activity, etc.). The app sharing board will be a moderated discussion platform and feed for participant interaction by posting healthy lifestyle practices through text, photographs and video to foster discussion on HTN management barriers/facilitators. The project team will post weekly to the sharing board on HTN-related topics to generate discussion among patients.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to test the hypertension (HTN) app-based intervention to see if it is more effective in improving uncontrolled HTN and HTN self-care among Africian-Americans from baseline to post-intervention (immediate, 3 months and 6 months post-intervention) as compared to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* African-American (AA) adults that are established patients at Neighborhood HealthSource in Minneapolis, Minnesota.
* Receives primary care (i.e., has designated primary care provider) at the partnering FQHCs and intent to continue care there for next 12 months
* African American race/ethnicity
* Men and women aged ≥18 years
* Uncontrolled HTN (defined as Stage 2 HTN with a BP ≥140/90 mmHg [as per 2017 American College of Cardiology/American Heart Association HTN Guidelines32] at most recent outpatient evaluation, with or without BP medications)
* Documented diagnosis of HTN in EHR
* At least 1 office visit at the partnering FQHCs in the prior year
* Smartphone ownership (supporting iOS or Android Systems)
* Active email address and willingness to utilize it throughout the study
* Basic Internet navigation skills (for example, can search for information on websites, open and send emails)
* Access to the Internet on at least a weekly basis (such as at home, a family member's or friend's home, church, library/community center, school/university, Internet café, etc.)?

Exclusion Criteria:

* Diagnosis of a serious medical condition or disability that would make participation difficult (i.e. visual or hearing impairment, mental disability that would preclude independent use of the app).
* No primary care provider at partnering FQHC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Absolute Change in Systolic Blood Pressure (BP) | Baseline, immediate post intervention
  Systolic BP (mmHg) will be measured as an average of 3 sitting readings with an oscillometric automated device during in-clinic health assessments.
HTN Self-Care as reported by H-SCALE(HTN Self-Care Activity Level Effects) | Baseline, immediate, 3 months, 6 months post intervention
  The H-SCALE is a 31-item instrument that assesses 6 HTN behavioral self-care activities recommended for optimal HTN management (BP medication adherence, weight loss/ideal body weight maintenance, adoption of a low-salt diet, regular physical activity for ≥30 minutes/day, limiting alcohol intake, and ceasing tobacco use).

SECONDARY OUTCOMES:
Proportion of subjects reaching BP control | Immediate, 3 months, 6 months post intervention
  Proportion of subjects reaching BP control (defined as meeting target BP of <140/90 mmHg)
Change in BP as assessed by home BP cuff measurements | Baseline, immediate post intervention
  BP (mmHg) will be measured 3 times per week during the 11-week intervention period using a home BP monitoring system. The 3 weekly measurements will be averaged and average weekly BP will be compared from baseline to immediate post intervention to determine the change in BP. This outcome is only evaluated in the intervention group as the control group will not undergo home BP cuff measurements.
CV Health Knowledge as measured by module assessment scores | Immediate post intervention
  Change in percentage correct scores (pre- and post- self-assessments) for each education module by patient and as a conglomerate (mean) for all patients.
Hypertension (HTN) Knowledge as assessed by 11-item questionnaire | Baseline, immediate post intervention
  HTN Knowledge will be assessed using a previously validated 11-item questionnaire which asks participants questions about the definition, prevention, management and complications of hypertension. Responses are record as true, false or uncertain to each question with true response receiving a score of 1 and false or uncertain responses receiving a score of 0. Total scores on the questionnaire range from 0-11 with higher scores reflecting better HTN knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess Brewer, M.D., M.P.H, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No